CLINICAL TRIAL: NCT01728922
Title: Dose-related Effects of Vitamin D3 on Immune Responses in Patients With Clinically Isolated Syndrome and Healthy Control Participants. An Exploratory Double Blind Placebo Randomised Controlled Study.
Brief Title: Dose-related Effects of Vitamin D3 on Immune Responses in Patients With Clinically Isolated Syndrome
Acronym: CISAVID
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University College Dublin (Other)
Collaborators: University of Dublin, Trinity College (Other); St Vincent's University Hospital, Ireland (Other)
Responsible Party: Principal Investigator, Professor Michael Hutchinson, Consultant Neurologist, Newman Clinical Research Professor, University College Dublin
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012CIS/VD/SVUH
Record Dates: First submitted 2012-11-08; First posted 2012-11-20 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Clinically Isolated Syndrome; Multiple Sclerosis
Keywords: Clinically isolated syndrome; Multiple sclerosis; Vitamin D; Immune response; CD4 T cell subsets; Cytokine
MeSH Terms: conditions — Multiple Sclerosis | interventions — Vitamin D

STUDY DESIGN:
Intervention Model Description: double-blind, dose ranging, two doses of vitamin D, randomised parallel groups with placebo arms in clinically isolated syndrome and heathy control participants
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: similar appearance of placebo and active drug
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Healthy control - 5,000 IU vitamin D (Active Comparator): 13 healthy controls will be administered 5,000 IU vitamin D. Primary outcome and safety outcome measures will be assessed.
  Interventions: Dietary Supplement: 5000IU vitamin D
- Healthy control - 10,000 IU vitamin D (Active Comparator): 13 healthy controls will be administered 10,000 IU vitamin D. Primary outcome and safety outcome measures will be assessed.
  Interventions: Dietary Supplement: 10000IU vitamin D
- CIS - placebo (Placebo Comparator): 15 patients will be administered placebo and all outcome measures will be assessed.
  Interventions: Other: Placebo
- CIS - 5,000 IU vitamin D (Active Comparator): 15 patients will be administered 5,000 IU vitamin D and all outcomes will be assessed.
  Interventions: Dietary Supplement: 5000IU vitamin D
- CIS - 10,000 IU vitamin D (Active Comparator): 15 patients will be administered 10,000 IU of vitamin D and all outcome measures assessed.
  Interventions: Dietary Supplement: 10000IU vitamin D
- Healthy control - placebo (Placebo Comparator): 13 control participants who will be administered placebo. These will be assessed for the primary outcome and safety outcomes only.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: 5000IU vitamin D — Vigantol Oil
  Other Names: Vigantol Oil
  Arms: CIS - 5,000 IU vitamin D; Healthy control - 5,000 IU vitamin D
Dietary Supplement: 10000IU vitamin D — Vigantol Oil
  Other Names: Vigantol Oil
  Arms: CIS - 10,000 IU vitamin D; Healthy control - 10,000 IU vitamin D
Other: Placebo — Placebo Oil
  Other Names: Placebo Oil
  Arms: CIS - placebo; Healthy control - placebo

SUMMARY:
The primary purpose of this study is to assess the immune response to vitamin D supplementation at two doses (5,000 IU and 10,000 IU daily) in both healthy controls and patients with clinically isolated syndrome compared to placebo. Secondary endpoints include (1) disease outcome in the clinically isolated syndrome in terms of clinical relapses and evidence of new lesions on MRI (McDonald's MS), 2) Safety of doses used

DETAILED DESCRIPTION:
Primary endpoint: To determine the effects of vitamin D supplementation at two doses a) 5,000 IU daily b) 10,000 IU daily compared to c) placebo a 24 weeks period on the change from baseline in frequency of CD4 T cell subsets and cytokine responses by peripheral blood mononuclear cells in 1) patients with the clinically isolated syndrome. 2) healthy control participants.

Secondary endpoints:

1. To determine whether there is a dose response effect of supplementation using 5,000 IU and 10,000 IU of vitamin D versus placebo over 24 weeks on the change from baseline in the frequency of CD4 T cell subsets and cytokine responses by PBMC in 1) patients with the clinically isolated syndrome (CIS) 2) healthy control participants
2. To establish whether there is a clinical response to vitamin D measured by a) change in the number of T2 lesions and Gadolinium enhancing lesions on MRI scanning at 24 weeks compared to baseline b) reduction in relapses over 24 weeks in treated (both 5,000 IU and 10,000 IU) CIS patients versus CIS patients receiving placebo.

ELIGIBILITY:
Inclusion Criteria: To be eligible for inclusion, each subject must meet each of the following criteria at Screening (Visit 1) and must continue to fulfil these criteria at Baseline (Visit 2).

* CIS: Patients with a clinically isolated syndrome with onset relapse within the previous three months and two or more than two asymptomatic T2 lesions on MRI brain scan.
* Aged 18-55yrs.
* Not receiving any disease modifying therapy.

Exclusion Criteria:

* Patients in whom any disease other than demyelination could explain their signs and symptoms.
* Participants with known disease of the parathyroids, a history of vitamin D intolerance, sarcoidosis, a history of hypercalcaemia of any cause.
* Participants with a baseline abnormality in serum urea, creatinine, calcium, parathormone.
* Participants on thiazide diuretics (hypercalcaemia risk).
* Patients with occurrence of a relapse less than six weeks prior to entry to study.
* Previous treatment with beta-interferons or glatiramer acetate or steroids in the last three months.
* Any previous treatment with mitoxantrone or other immunosuppressant.
* Participants already taking supplemental vitamin D.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2012-11-06 (Actual); Primary Completion 2015-06-05 (Actual); Study Completion 2016-06-05 (Actual)

PRIMARY OUTCOMES:
The effects of two doses of vitamin D and placebo therapy on the change in the frequency of CD4 T cell subsets and cytokine responses of PBMC over 24 weeks of therapy from baseline. | This outcome measure will be assessed at baseline and at 24 weeks.
  A number of measures will be examined in particular IL-10 production and the frequency of Th17 cells.

SECONDARY OUTCOMES:
The number of new T2 and gadolinium enhancing lesions compared to baseline amongst the study group. | Baseline and 24 weeks
  The MRI out-come measure will assess the a) number of Gadolinium enhancing lesions b) the number of new and enlarging T2 lesions c) the combined unique lesion count (new and enlarging T2 lesions plus Gadolinium enhancing lesions) after 24 weeks of therapy in the three arms, 5000IU, 10,000IU vitamin D and placebo . Mean and median new T2 and gadolinium-enhancing lesions at 24 weeks (end of the trial) will be compared for each treatment allocation group. In addition the mean and median number of new T2 lesions plus gadolinium enhancing lesions in all the CIS patients on vitamin D will be compared to the mean and median in the placebo group.
Relapse occurrence in the CIS patients during 24 weeks of the trial | At each clinic visit or as the need arises.
  Relapse occurrence in the CIS patients during 24 weeks of the trial;(i) annualised relapse rates (ARR), (ii) percentage of patients free from relapses and (iii) time to first relapse will be compared for each treatment allocation group. In addition the same relapse measures will be applied to both vitamin D treated groups combined and compared to those in the placebo group.
The percentage of CIS patients in each treatment arm free from any evidence of disease activity (No relapses, no new T2 lesions, no gadolinium enhancing lesions). | At 24 weeks.

OTHER OUTCOMES:
Serum calcium | Every 4 weeks for 24 weeks
  a measure of calcium homeostasis
Number of participants with adverse events as a measure of safety and tolerability of vitamin D in doses of 5,000IU and 10,000IU daily | four weekly assessments over 24 weeks
serum urea | 4 weekly over 24 weeks
  a measure of renal function
serum creatinine | 4 weekly over 24 weeks
  a measure of renal function
serum 25(OH)D levels | 4 weekly over 24 weeks
  a measure of response to oral dosing and adherence to therapy.
serum parathormone (iPTH) | 4 weekly over 24 weeks
  a measure of parathyroid function

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hutchinson, MB, FRCP, Principal Investigator — St Vincent's University Hospital, Ireland
Locations (1):
- St Vincent's University Hospital, Dublin, Dublin 4, Ireland

IPD SHARING:
Plan to Share IPD: Yes
all demographic details and outcome measures may be obtained directly from the PI by e-mail

REFERENCES:
- [Derived] O'Connell K, Kelly S, Kinsella K, Jordan S, Kenny O, Murphy D, Heffernan E, O'Laoide R, O'Shea D, McKenna C, Cassidy L, Fletcher J, Walsh C, Brady J, McGuigan C, Tubridy N, Hutchinson M. Dose-related effects of vitamin D on immune responses in patients with clinically isolated syndrome and healthy control participants: study protocol for an exploratory randomized double- blind placebo-controlled trial. Trials. 2013 Aug 27;14:272. doi: 10.1186/1745-6215-14-272. PMID 23981773